CLINICAL TRIAL: NCT03328091
Title: Genetic Counseling Processes and Outcomes Among Males With Prostate Cancer (ProGen)
Acronym: ProGen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Huma Rana, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-409
Record Dates: First submitted 2017-10-25; First posted 2017-11-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Genetics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional pre-test genetic counseling (Active Comparator): * In-person consultation with licensed genetic counselor at the Center for Cancer Genetics and Prevention before genetic testing
  * Participant is given a pamphlet introducing prostate cancer genes, genetic testing
  * Participant is sent electronic family history tool
  * Participant is given the "Genetic Testing Information for Decision Making" packet. After the genetic counseling session, patient is asked if they would like to proceed with genetic testing.
  Interventions: Other: Traditional pre-test genetic counseling
- Pre-test video education (Experimental): * Participant is given a pamphlet that describes the basics of prostate cancer genes, genetic testing
  * Participant is sent electronic family history tool
  * Participant is approached in clinic by research staff at a pre-planned time
  * The patient is given the "Genetic Testing Information for Decision Making" packet
  * The pre-test video education is a short video. Information will be provided about the basics of genetics and mutations, the potential benefits, risks, and limitations of genetic testing, and the possible results the participant may receive
  Interventions: Other: Pre-test video education

INTERVENTIONS:
Other: Traditional pre-test genetic counseling — Participant meets with a genetic counselor at the Center for Cancer Genetics and Prevention and traditional pre-test cancer genetic counseling is provided
  Arms: Traditional pre-test genetic counseling
Other: Pre-test video education — The video is designed to mirror the educational components of a traditional genetic counseling visit
  Arms: Pre-test video education

SUMMARY:
This randomized controlled trial aims to evaluate the impact of pre-test video education and post-test genetic counseling as compared to in-person pre-test genetic counseling in males with advanced prostate cancer.

DETAILED DESCRIPTION:
Participants will be randomized to either pre-test video education and post-test genetic counseling or in-person pre-test genetic counseling. Outcomes evaluated are: prevalence of germline mutations, uptake of genetic testing, satisfaction with testing, knowledge of multi-gene panels, distress, result disclosure to relatives, and the impact on personal or family medical care. Through this study, the investigators will learn about the inherited causes of prostate cancer, and how and when genetic testing should be offered to this population.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic prostate cancer (hormone-sensitive, de novo, or castration resistant)
* Localized prostate cancer with Gleason score ≥8
* Rising PSA after prostatectomy or radiation with PSA doubling time ≤ 6 months
* Persistent PSA after prostatectomy for PSA ≥ 0.2 ng/mL observed in testing at least 1 week apart
* Prostate cancer diagnosed at age ≤ 55 years
* Prostate cancer and a personal history of prior malignancy that does not include non-melanoma skin cancer or superficial bladder cancer.
* Prostate cancer diagnosis (any grade/stage) or prostate biopsy with high grade PIN or small acinar proliferation and a family history potentially indicating a germline mutation (e.g. breast cancer diagnosed at age ≤ 50, ovarian, pancreatic, uterine, colorectal, prostate cancer or sarcoma, in one or more first or second-degree relatives)

Exclusion Criteria:

* Previous cancer genetic testing or counseling, or prior germline multigene panel testing. Previous tumor sequencing is acceptable if no genetic counseling took place.
* Localized prostate cancer previously treated and in remission for > 2 years unless family history potentially indicates a germline mutation.
* Active hematologic malignancy (e.g. CLL)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of germline mutations in males with prostate cancer | 2 years
  The proportion of participants who test positive for pathogenic or likely pathogenic variants

SECONDARY OUTCOMES:
Genetic testing uptake | 2 years
  The proportion of participants who consent to genetic testing in the pre-test video education arm
Secondary or other primary (non-prostate) malignancies | 2 years
  Assessed by chart review. Participants with positive genetic test results will fill out the "Positive Test Results" Survey to report any additional cancer diagnoses.
Genetic testing satisfaction score | at time of post-counseling/video pre-result disclosure and at 1 month post-result disclosure
  A validated survey of participants' satisfaction with the genetic counseling and testing process will be used. For the survey at the time of post-counseling, the survey for the video education arm consists of 8 questions and the genetic counseling arm contains an additional question about perceived length of the visit. The parameters for measurement are "disagree strongly", "disagree", "neither agree or disagree", "agree", and "agree strongly". At the time of 1 month post-result disclosure, an additional set of 5 questions will be added. Four of these five questions will be evaluated using the previously described parameters. The remaining question will be answered by the response options: "yes", "no", or "I did not get the packet". Survey responses will be re-coded on a numerical scale consistent with the standard Likert scale.
Multidimensional Impact of Cancer Risk Assessment score and subscales | 1 and 4 months post-result disclosure
  MICRA is a widely used validated 25-item measure that assesses psychosocial consequences associated with genetic testing for cancer. Section 1 contains 3 sub-scales: the Positive sub-scale (4 items), the Distress sub-scale (6 items), and the Uncertainty sub-scale (9 items) and two other items that do not fit into either sub-scale. Section 2 contains two items for participants who have children. Section 3 contains 2 items for participants who have/have had cancer. Responses are indicated on a 4 point scale for experiences in the past week. A higher score in the sub-scales or total scale indicated greater distress. The positive sub-scale is reverse scored to reflect this.
Knowledge of multigene panel testing score | 4 months post-result disclosure
  A 24 item investigator-developed knowledge scale applicable to this population was developed through an expert panel and in-depth patient cognitive interviews to determine if participants are able to recall key core components about multi-gene panel testing. Each item provides three choice answers: "agree", "disagree", or "I don't know". Knowledge will be scored on the number of "correct" responses where higher correct responses represents more knowledge of multigene panel testing.
Family communication for those who tested positive for a genetic mutation | 1 and 4 months post-result disclosure
  For those participants who have tested positive for a mutation, 5 items will be asked pertaining to disclosure of genetic testing results to relatives that are derived from previous literature.
Intent to disclose genetic test results | pre-result disclosure
  Three items will assess participants' intentions to disclose genetic testing results.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Q Rana, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rana HQ, Stopfer JE, Weitz M, Kipnis L, Koeller DR, Culver S, Mercado J, Gelman RS, Underhill-Blazey M, McGregor BA, Sweeney CJ, Petrucelli N, Kokenakes C, Pirzadeh-Miller S, Reys B, Frazier A, Knechtl A, Fateh S, Vatnick DR, Silver R, Kilbridge KE, Pomerantz MM, Wei XX, Choudhury AD, Sonpavde GP, Kozyreva O, Lathan C, Horton C, Dolinsky JS, Heath EI, Ross TS, Courtney KD, Garber JE, Taplin ME. Pretest Video Education Versus Genetic Counseling for Patients With Prostate Cancer: ProGen, A Multisite Randomized Controlled Trial. JCO Oncol Pract. 2023 Nov;19(11):1069-1079. doi: 10.1200/OP.23.00007. Epub 2023 Sep 21. PMID 37733980
- [Derived] Berchuck JE, Boiarsky D, Silver R, Sunkara R, McClure HM, Tsai HK, Siegmund S, Tewari AK, Nowak JA, Lindeman NI, Rana HQ, Choudhury AD, Pomerantz MM, Freedman ML, Van Allen EM, Taplin ME. Addition of Germline Testing to Tumor-Only Sequencing Improves Detection of Pathogenic Germline Variants in Men With Advanced Prostate Cancer. JCO Precis Oncol. 2022 Aug;6:e2200329. doi: 10.1200/PO.22.00329. PMID 36103646